CLINICAL TRIAL: NCT03680573
Title: The Effect of Antioxidants on Skin Blood Flow-BH4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Responsible Party: Principal Investigator, Matthew Brothers, Associate Professor, The University of Texas at Arlington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-0842
Record Dates: First submitted 2018-09-17; First posted 2018-09-21 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factor; Vasoconstriction
Keywords: Racial Differences; Oxidative Stress
MeSH Terms: conditions — Cardiovascular Diseases | interventions — acetovanillone; Allopurinol; NG-Nitroarginine Methyl Ester; Nitroprusside; Erythrocyte Indices

STUDY DESIGN:
Intervention Model Description: Each subject has one control site and three experimental sites concurrently tested within the same study using intradermal microdialysis on the dorsal forearm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Control- Lactated Ringers (Active Comparator): This site will serve as the control site and will receive lactated Ringer's (saline solution) at an infusion rate of 2 µl/min.
  Interventions: Drug: Control: Lacated Ringers; Drug: NG Nitro L Arginine Methyl Ester; Drug: Sodium Nitroprusside; Drug: Acetyl-ß-methylcholine chloride
- Apocynin (1-(4-Hydroxy-3-methoxyphenyl)ethanone) (Experimental): This site will receive 100 µM apocynin (1-(4-Hydroxy-3-methoxyphenyl)ethanone) at an infusion rate of 2 µl/min.
  Interventions: Drug: Apocynin; Drug: NG Nitro L Arginine Methyl Ester; Drug: Sodium Nitroprusside; Drug: Acetyl-ß-methylcholine chloride
- Allopurinol (1H-pyrazolo[3,4-d]pyrimidin-4(2H)-one) (Experimental): This site will receive 10 µM allopurinol (1H-pyrazolo[3,4-d]pyrimidin-4(2H)-one)at an infusion rate of 2 µl/min.
  Interventions: Drug: Allopurinol; Drug: NG Nitro L Arginine Methyl Ester; Drug: Sodium Nitroprusside; Drug: Acetyl-ß-methylcholine chloride
- BH4 ((6R)-5,6,7,8-Tetrahydrobiopterin dihydrochloride) (Experimental): This site will receive 10 mM (6R)-5,6,7,8-Tetrahydrobiopterin dihydrochloride (BH4) at an infusion rate of 2 µl/min.
  Interventions: Drug: BH4; Drug: NG Nitro L Arginine Methyl Ester; Drug: Sodium Nitroprusside; Drug: Acetyl-ß-methylcholine chloride

INTERVENTIONS:
Drug: Control: Lacated Ringers — This site will serve as the control site
  Arms: Control- Lactated Ringers
Drug: Apocynin — This site will be used to inhibit NADPH oxidase and subsequent production of superoxide.
  Arms: Apocynin (1-(4-Hydroxy-3-methoxyphenyl)ethanone)
Drug: Allopurinol — This site will be use to inhibit xanthine oxidase and subsequent production of superoxide.
  Arms: Allopurinol (1H-pyrazolo[3,4-d]pyrimidin-4(2H)-one)
Drug: BH4 — This site will be use to locally supplement BH4.
  Arms: BH4 ((6R)-5,6,7,8-Tetrahydrobiopterin dihydrochloride)
Drug: NG Nitro L Arginine Methyl Ester — L-Name is a NOS inhibitor that is administered to each site to allow for the quantification of NO contribution to vasodilation. The infusion rate will be 2 µl/min
  Other Names: L-Name
Drug: Sodium Nitroprusside — SNP will be perfused through each site to induce maximal vasodilation. The infusion rate will be 2 µl/min
  Other Names: SNP
Drug: Acetyl-ß-methylcholine chloride — Mch is an acetylcholine analog that causes endothelial dependent vasodilation primarily through stimulation of NO production.
  Other Names: Mch

SUMMARY:
The goal of this study is to examine possible mechanisms of heightened vasoconstriction in Black/African American men and women as possible links to the elevated prevalence of cardiovascular dysfunction and disease. The main targets in this study are sources of oxidative stress

DETAILED DESCRIPTION:
African Americans (AA) not only have a higher prevalence of hypertension but the severity of the cardiovascular complications related to this condition are greater in this population relative to other populations. While the underlying causes of this elevated risk are multifactorial, vascular dysfunction (i.e. impaired vasodilation and/or augmented vasoconstriction) is believed to be a key contributing factor. The investigators have recently observed (UTA IRB 2016-0268) that the small blood vessels in the skin (the cutaneous microvasculature) in AA, but otherwise healthy individuals, have an impaired blood flow response in the cutaneous circulation to local heating when compared to age, body mass index (BMI), and gender, matched Caucasians (CA). This blunted response is abolished in AA when the sites are pre-treated with either Allopurinol or Apocynin which block the production of xanthine oxidase and NADPH oxidase, respectively. In addition, Tetrahydrobiopterin (BH4) is critically involved in vascular function. BH4 is a cofactor involved in the conversion of L-Arginine into the potent vasodilator nitric oxide (NO) by the enzyme endothelial nitric oxide synthase (eNOS). Reduced bioavailable BH4 leads to elevated oxidative stress and thus impaired vascular function.

In addition to local heating another commonly utilized research approach to assess microcirculatory vascular function is via local infusion of the potent vasodilator methacholine (Mch). Mch is an acetylcholine analog that causes endothelial dependent vasodilation primarily through stimulation of NO production. Much like the local heating data mentioned above, our laboratory (data collected while at UT Austin) has demonstrated a blunted response to Mch in AA relative to CA. However, the role of xanthine oxidase, NADPH oxidase, and BH4 in this blunted response remains unknown.

ELIGIBILITY:
Inclusion Criteria:

* Individuals (ages 18-35, both genders) will be recruited from the greater Arlington area to participate in the study.
* Must self-report both parents as either African American or Caucasian American.

Exclusion Criteria:

* Individuals who have donated more than 550 ml of blood within the past 8 weeks will not have blood drawn from them in this protocol. However, if they remain interested in the study, and otherwise meet the inclusion criteria, than we may still opt to proceed with data collection.
* Individuals with cardiovascular, neurological, and/or metabolic illnesses will be excluded from participating as well as individuals with a history of various diseases of the microvasculature including Reynaud's disease, cold-induced urticaria, cryoglobulinemia, etc.
* Subjects currently taking any prescription medications and individuals with a body mass index about 30 kg/m2) will be excluded.
* Pregnant subjects and children (i.e. younger than 18) will not be recruited for the study. Eligible females will be scheduled for days 2-7 of their menstrual cycle to account for hormonal effects on blood flow. A regular menstrual cycle is required to identify and schedule the study for the low hormone period, therefore females who lack a regular cycle will be excluded from the study. Females currently taking birth control are eligible, as long as they can be scheduled during a low-hormone "placebo" week. If their hormone do not contain a placebo week than these individuals will not be eligible for data collection. Females who are breast-feeding will also be eligible as there are no systemic or lasting effects of the proposed vasoactive agents.
* Given that smoking can affect the peripheral vasculature, current smokers and individuals who regularly smoked (>1 pack per two weeks) within the prior 2 years will be excluded

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-05-05 (Actual); Study Completion 2018-05-05 (Actual)

PRIMARY OUTCOMES:
Blood Flow Response to the Administration of Methacholine (Mch) before and after Infusions of Vasoactive Drugs using Intradermal Microdialysis and Laser Doppler Fluxmetry | Through study completion, an average of 1 Year
  To establish impaired blood flow response to local administration of Mch in African American relative to Caucasians. Mch will be administered using intradermal microdialysis in separate doses while the skin blood flux response will be determined using laser Doppler fluxmetry. All changes in flux will be normalized and reported as a percentage of maximal flux. The role of oxidative stress and low nitric oxide synthase cofactors will be assessed using infusions of apocynin/allopurinol and tetrahydrobiopterin (BH4), respectively. These infusions will be given after the first infusion of Mch and before the second infusion of Mch to determine how Mch responsiveness changes with these vasoactive drugs.

CONTACTS AND LOCATIONS:
Locations (1):
- Engineering Research Building, Arlington, Texas, United States

IPD SHARING:
Plan to Share IPD: No